CLINICAL TRIAL: NCT02715687
Title: Treatment of Postoperative Atrial Fibrillation - Comparison of Amiodarone and Placebo.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ziv Beckerman MD, MD, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AF Treatment
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Will receive 30 days treatment with oral placebo of 200mg
  Interventions: Drug: Placebo
- Interventional (Active Comparator): Will receive 30 days treatment with oral Amiodarone of 200mg
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Amiodarone — Will receive 30 days treatment with oral amniodarone of 200mg
  Other Names: amiodacore
  Arms: Interventional
Drug: Placebo — Will receive 30 days treatment with oral placebo of 200mg
  Arms: Placebo

SUMMARY:
Post-operative atrial fibrillation (POAF) is the most common complication encountered after cardiac surgery; reports show POAF to occur in ~ 35% of patients after CABG. Prophylactic use amiodarone was found to be effective, however, due to serious extracardiac adverse effects therapy is probably appropriate just for patients at high risk for POAF.

the common practice for management of POAF is treatment with intravenous Amiodarone until return to sinus rhythm, following which the drug is given orally. Our protocol involves continued treatment with amiodarone for 30 day post-discharge from the hospital in a dose of 200mg per day.

This protocol is a common practice in many cardiac surgical departments worldwide, nevertheless, it is not evidence-based protocol and it was never examined as such.

This study is a randomized placebo controlled trial, to evaluate the requirement for post-discharge treatment with oral Amiodarone.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most widespread complication encountered after cardiac surgery, associated with prolonged hospitalization, morbidity, mortality, and an annual cost of more than $1 billion to the American healthcare system.

AF has been reported to predict postoperative stroke, congestive heart failure, and late AF among patients undergoing mitral valve surgery. Postoperative AF (POAF) occurs in 62% of patients undergoing combined aortic valve and coronary artery bypass graft (CABG) surgery, in 49% of patients undergoing aortic valve surgery alone, in 42% of patients undergoing mitral valve surgery, and in 32% of patients undergoing CABG surgery alone. These figures are expected to rise in the future, given that the patients undergoing cardiac surgery are getting elder and that the incidence of AF in the general population is markedly age-dependent.

POAF peak incidence occurs on the 2nd and 3rd postoperative days (PODs). Seventy percent of patients develop this arrhythmia before the end of the 4th POD and 94% before the end of the 6th. Although generally well-tolerated and seen as a temporary problem related to surgery, POAF can be life-threatening, particularly in elderly patients and those with left ventricular dysfunction.

Recent guidelines for the prevention and management of POAF were jointly published in 2006 by the American College of Cardiology, the American Heart Association (AHA), and the European Society of Cardiology. These guidelines recommended (i) preoperative treatment with an oral beta-blocker drug for prevention of POAF as a class IA indication, and (ii) preoperative administration of amiodarone for patients at a high risk for POAF as a class IIA indication.

Amiodarone is associated with several complications, both cardiac, and extracardiac; among the cardiac complications, it is predominantly related to increased risk of bradycardia and hypotension, particularly when (i) administered intravenously, (ii) using average daily doses exceeding 1 g, and (iii) initiating prophylaxis during the postoperative period.45 Among the most severe extracardiac complications, amiodarone is associated with thyroid toxicity, lung fibrosis, and corneal damage, which may be aggravated by the drug's delayed onset of action (2 - 3 days) and long elimination half-life time (up to 6 months).

Currently the common practice for management of POAF is treatment with intravenous Amiodarone until return to sinus rhythm, following which the drug is given orally. Our protocol involves continued treatment with amiodarone for 30 day post-discharge from the hospital in a dose of 200mg per day.

This protocol is a common practice in many cardiac surgical departments worldwide, nevertheless, it is not evidence-based protocol and it was never examined as such.

This study is a randomized placebo controlled trial, to evaluate the requirement for post-discharge treatment with oral Amiodarone.

ELIGIBILITY:
Inclusion Criteria:

* All post-cardiac surgery patients who developed a hemodynamically stable postoperative atrial fibrillation and returned to sinus rhythm with intravenous amiodarone tretament.

Exclusion Criteria:

* Post-cardiac surgery patients who developed a non- hemodynamically stable postoperative atrial fibrillation.
* Patients with chronic and/or paroxysmal atrial fibrillation and/or known other cardiac arrhythmia or conduction disturbance.
* Patients with pacemakers.
* Patients with lactose intolerance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation | 30 days after discharge
  Post-discharge monitoring with a continous loop-recorder type of ECG monitoring device named "CardioR" will be provided for all participants. The device will continuously record and transmit ECG monitoring to a dedicated monitoring company. All arrhythmias will be recorded and reported.

SECONDARY OUTCOMES:
Post-discharge return to admission | 30 days after discharge
  Any return to admission will be recorded and reported.

IPD SHARING:
Plan to Share IPD: Undecided